CLINICAL TRIAL: NCT00981851
Title: A Hazardous Combination of Cigarette Smoking and Bronchodilation in Chronic Obstructive Pulmonary Disease
Brief Title: Interaction in Chronic Obstructive Pulmonary Disease Experiment
Acronym: ICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: TRJ Schermer, PhD, Radboud University Nijmegen Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: RvB08.066.51196/GE
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Cardiovascular Disease; Smoking; Bronchodilation
Keywords: intervention study; interaction; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Smoking | interventions — Tiotropium Bromide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- beta 2 agonist + anticholinergic aerosol (Active Comparator)
  Interventions: Drug: Tiotropium (Spiriva) + Salbutamol (Ventolin)
- placebo inhalation (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tiotropium (Spiriva) + Salbutamol (Ventolin) — 1 time inhalation of 5 mcg of Tiotropium bromide by Respimat and 400 mcg of Salbutamol by Volume Spacer. cigarette smoking
  Other Names: Spiriva Respimat; Ventolin Aerosol
  Arms: beta 2 agonist + anticholinergic aerosol
Drug: placebo — 1 time inhalation of placebo with the amount of puffs similar to the active comparator. cigarette smoking
  Other Names: Ventolin placebo and Spiriva placebo
  Arms: placebo inhalation

SUMMARY:
The final purpose of this study is to determine whether bronchodilation and cigarette smoking in Chronic Obstructive Pulmonary Disease (COPD) patients interact, resulting in an increase of cardiovascular disease. The aim of this part of the study is to demonstrate the basic mechanism: Does increased respiratory function after administration of a bronchodilator in patients with COPD lead to elevated pulmonary retention of the harmful compounds in inhaled cigarette smoke and to short-term biological effects associated with cardiovascular disease?

DETAILED DESCRIPTION:
COPD currently is one of the most frequent diseases. In more than 80% of COPD patients, the disease is caused by smoking. About half of the COPD patients are active smokers, although smoking is also the most important prognostic factor. Also, smoking is an important cause as well as an important prognostic factor in cardiovascular disease. The corner stone of medical treatment in COPD is bronchodilation; more than half of the patients use a long-acting bronchodilator. An increase of the pathogenic effect of smoking by an increased lung function after bronchodilation is likely though, since more pathogenic particles would penetrate the lung. We hypothesize that bronchodilators increase cardiovascular disease in COPD patients who smoke.

In order to demonstrate the basic mechanism of our hypothesis, COPD patients receive a bronchodilator at one time and a placebo at another time, preceded and followed by cigarette smoking during one hour as by a strict time schedule. Smoke retention, lung function and blood biomarkers are repeatedly measured.

ELIGIBILITY:
Inclusion Criteria:

* COPD Gold stage II-III (FEV1/FVC<0,70 and FEV1 30-80% of predicted value).
* Current cigarette smoking (at the time of performing the study).
* Willing to provide written informed consent.
* Refrain from smoking and bronchodilators > 8 hours (depends on treatment) before the test.
* Registered in one of the recruitment institutes.

Exclusion Criteria:

* COPD gold stage I or IV.
* Asthmatic component: History of asthma, present asthma by complaints, eosinophilia or reversibility ≥ 10% of predicted.
* Unable to communicate.
* Physically unable to perform any of the tests.
* Non-COPD respiratory disorders.
* Previous lung-volume reduction surgery and/or lung transplantation.
* Evidence of alcohol, drug or solvent abuse.
* Known α-1 antitrypsin deficiency.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
cigarette smoke retention | retention measurement is during smoking. smoking is 1 cigarette before and 1 cigarette 45 minutes after medication inhalation for each arm. 1 week between arms

SECONDARY OUTCOMES:
(hs)CRP | 3 times within 2 hours for each arm
fibrinogen | 3 times within 2 hours for each arm
respiratory function | at baseline and repeatedly around medication inhalation for 1.5 hours
smoking pattern: smoke inhalation and smoke exhalation time and volume | during smoking cigarettes: twice for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Tjard RJ Schermer, PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (2):
- Netherlands (2):
  - University Center for Chronic Diseases Dekkerswald, Groesbeek
  - Primary care, general practitioners, Nijmegen

REFERENCES:
- [Derived] van Dijk WD, Heijdra Y, Lenders JW, Klerx W, Akkermans R, van der Pouw A, van Weel C, Scheepers PT, Schermer TR. Cigarette smoke retention and bronchodilation in patients with COPD. A controlled randomized trial. Respir Med. 2013 Jan;107(1):112-9. doi: 10.1016/j.rmed.2012.09.019. Epub 2012 Oct 12. PMID 23069326
- [Derived] van Dijk WD, Scheepers PT, Cremers R, Lenders JW, Klerx W, van Weel C, Schermer TR, Heijdra Y. A method to study the effect of bronchodilators on smoke retention in COPD patients: study protocol for a randomized controlled trial. Trials. 2011 Feb 10;12:37. doi: 10.1186/1745-6215-12-37. PMID 21310040